CLINICAL TRIAL: NCT07274514
Title: Effects of Immersive Virtual Reality on Balance of Parkinson's Disease
Brief Title: Virtual Reality on Balance of Parkinson's Disease
Acronym: RVI-PD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Sanitaria Aragón (Other)
Collaborators: Universidad San Jorge (Other); Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Sandra Calvo Carrión, PhD, Instituto de Investigación Sanitaria Aragón
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UZ-USJ-PD
Record Dates: First submitted 2025-08-21; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-10

CONDITIONS: Parkinson Disease (PD); Immersive Virtual Reality; Physical Therapy
Keywords: Immersive Virtual Reality; Balance; Physical Therapy; Quality of life; Gait; Strength; parkinson's disease; virtual reality
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Single-blind randomized clinical trial with two parallel interventions
Who Masked: Outcomes Assessor
Masking Description: Single Blind (Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group. Immersive Virtual Reality Rehabilitation Program (Experimental): The participants in the experimental group will receive a immersive virtual reality rehabilitation program to improve static and dynamic balance and quality of life.
  Interventions: Other: Immersive Virtual Reality Program
- Control Group. Standard Rehabilitation Program (Active Comparator): The participants in the control group will receive a standard physical therapy rehabilitation program to improve static and dynamic balance and quality of life
  Interventions: Other: Standard Rehabilitation Program

INTERVENTIONS:
Other: Immersive Virtual Reality Program — The participants in the intervention group will receive a Immersive Virtual Reality Rehabilitation Program to improve static and dynamic balance and quality of life
  Arms: Intervention Group. Immersive Virtual Reality Rehabilitation Program
Other: Standard Rehabilitation Program — The participants in the control group will receive a Standard Physical Therapy Rehabilitation Program to improve static and dynamic balance and quality of life
  Arms: Control Group. Standard Rehabilitation Program

SUMMARY:
This study, titled: Effectiveness of immersive virtual reality on balance in people with Parkinson's disease. Is a randomized clinical trial conducted at Zaragoza Parkinson's Association in Spain. It aims to evaluate the effectiveness of a immersive virtual reality program in enhancing balance for patients with Parkinson.s disease (PD). PD is a neurodegenerative disease that has a major impact on patients' balance and gait, affecting their quality of life. Physical rehabilitation is crucial for maintaining and improving balance, and immersive virtual reality promises to be an alternative for improving outcomes in patients with PD.

DETAILED DESCRIPTION:
Study Backgroud and Rationale: Parkinson's disease (PD) is one of the most common neurogenerative disease. Parkinson's disease is one of the most common neurodegenerative diseases. Patients suffering from it present a series of motor symptoms, including resting tremors, hyperresistance, bradykinesia, postural instability, and gait disturbances. Postural instability leads to an increase in the number of falls, which leads to greater dependence and social isolation, resulting in a reduced quality of life. Usual physical therapy techniques show an improvement in the motor skills of people with PD; however, their effectiveness is sometimes limited by patient adherence. Objective: The primary objective of this study is to determine whether the Immersive Virtual Reality (IVR) program rehabilitation can improve the balance of people with PD by Mini-Balance Systems Test (Mini-BESTest). Secondary objectives included assessing changes in gait speed, lower limbs strength, functional mobility, quality of life, adherence to the treatment and the possible occurrence of adverse symptoms during the use of IVR. Study Design: This is a single-blind, randomized clinical trial. Fifty patients with PD will be recruited and randomly assigned to either the control group, wich will receive balance conventional physiotherapy rehabilitation thought or the intervention group, wich will receive a IVR program rehabilitation. Both groups will undergo a comprehensive rehabilitation program that will include: active mobility exercises, strength exercises for the main antigravity muscles, and active stretching of the main muscles of the posterior chain. Methodology: There will be eight 40-minute sessions over four weeks. The first 20 minutes will be the same for both groups, while the second part of the session will vary between the control group (standard physical therapy) and the intervention group (IVR).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PD confirmed by a neurologist
* Age between 55 and 90 years
* Hoehn & Yahr Scale score of 1 to 4
* Cognitive level of 24 or higher on the Mini Mental Examination Test
* Ability to stand upright without assistance

Exclusion Criteria:

* Visual or auditory impairments that could interfere with the perception of information or trigger dizziness or epilepsy
* Musculoskeletal conditions that hinder or prevent the execution of exercises or the ability to maintain a standing position for at least 20 minutes
* Psychiatric disorders such as moderate or severe depression diagnosed in the last year and impulse control disorders diagnosed in the last year
* Score of 20 points on the Simulator Sickness Questionnaire (SSQ scale), indicating the presence of severe adverse symptoms

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-02-05 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Balance-Mini-Balance Systems Test (Mini-BESTest) | Balance will be assessed at three time points: pre-intervention (M0), the day post-intervention (M1), and 90 days post-intervention (M2).
  The primary outcome is the improvement in balnace, which will be evaluated using the Mini-Balance Systems Test (Mini-BESTest). This test assesses static and dynamic balance disorders and determines the risk of falling by evaluating 14 items divided into 4 categories: anticipatory, reactive postural control, sensory orientation and dynamic gait. recovery.static and dynamic balance disorders and determines the risk of falling

SECONDARY OUTCOMES:
Gait speed-10-Meter Walk Test (10MWT) | Gait speed will be assessed at three time points: pre-intervention (M0), the day post-intervention (M1), and 90 days post-intervention (M2).
  Evaluate improvements in gait speed using the 10 meters walk test (10=MWT). The aim is to determine whether the immersive virtual reality program can enhance gait speed as compared to the usual physiotherapy approach.
Lower Limb Muscle Strength - 30 seconds Sit to Stand Test (30 CST) | Lower Limb Muscle Strength will be assessed at three time points: pre-intervention (M0), the day post-intervention (M1), and 90 days post-intervention (M2).
  Evaluate lower limb muscle strength using the 30 seconds sit-to-stand test (30CST). This assessment will provide data on the effectiveness of the immersive virtual reality program in improving lower extremity muscle strength
Functional mobility during walking-Time up and Go (TUG) | Balance will be assessed at three time points: pre-intervention (M0), the day post-intervention (M1), and 90 days post-intervention (M2).
  Assess the functional mobility during walking, as well as the risk of falling
Functional mobility performing a dual task-Time Up & Go Dual Task (TUG-DT): | Functional mobility performing a dual task will be assessed at three time points: pre-intervention (M0), the day post-intervention (M1), and 90 days post-intervention (M2).
  Asses functional mobility during walking, as well as the risk of falling while performing a dual task with Time Up and Go Dual Task (TUG-DT)
Quality of life- Parkinson Disease Questionnaire-39 (PDQ-39 | Quality of life will be assessed at three time points: pre-intervention (M0), the day post-intervention (M1), and 90 days post-intervention (M2).
  Assess health-related quality of life in people with PD. This self-administered questionnaire consists of 39 items, divided into eight dimensions (mobility, activities of daily living,emotional well-being,stigma, social support, cognition, comunication, bodily discomfort.
Adverse symptoms- Simulator Sickness Questionnaire (SSQ) | Through intervention completion, an average of 1 month.
  Assess the occurrence of adverse symptoms during the Immersive Virtual Reality Program using the Simulator Sickness Questionnaire (SSQ). This questionnaire consists of 16 items divided into three sections: Oculomotor Function, Nausea, and Disorientation.
Adherence to the Immersive Virtual reality program | Through intervention completion, an average of 1 month.
  Evaluate compliance with the immersive virtual reality program by monitoring the percentage of sessions completed by participants. The compliance rate will be calculated as the number of sessions completed relative to the total number of program sessions.
Satisfaction with Immersive Virtual Reality Program | Satisfaction with Immersive Virtual Realiity program will be assessed at two time points: the day post-intervention (M1), and 90 days post-intervention (M2).
  Evaluate participant satisfaction with the immersive virtual reality program using a standardized ad hoc questionnaire on a 5- point Likert scale, scored of 1 to 5, with higher scores indicating greater satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Calvo, PhD, Principal Investigator — Universidad de Zaragoza
Locations (1):
- Asociación de Parkinson de Aragón, Zaragoza, Spain